CLINICAL TRIAL: NCT03494179
Title: A Multicenter, Open-label Study to Evaluate the Safety and Efficacy of ICP-022 in Patients With Relapsed/Refractory Mantle Cell Lymphoma (MCL)
Brief Title: A Study to Evaluate ICP-022 in Patients With R/R Mantle Cell Lymphoma (MCL)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00102
Record Dates: First submitted 2018-03-19; First posted 2018-04-11 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Dose of ICP-022 (Experimental): Two regimens of ICP-022 (High dose QD and low dose BID) are designed for study Part I to determine RP2D which will be used in Part II to further evaluate the preliminary anti-tumor effects of ICP-022 in Chinese subjects with R/R MCL.
  Interventions: Drug: ICP-022
- Low Dose of ICP-022 (Experimental): Two regimens of ICP-022 (High dose QD and low dose BID) are designed for study Part I to determine RP2D which will be used in Part II to further evaluate the preliminary anti-tumor effects of ICP-022 in Chinese subjects with R/R MCL.
  Interventions: Drug: ICP-022

INTERVENTIONS:
Drug: ICP-022 — The drug product is a white, round, uncoated tablet.

SUMMARY:
The phase I/II clinical study is to investigate the safety, tolerability and pharmacokinetics/ pharmacodynamics of ICP-022.

DETAILED DESCRIPTION:
Part I: PK/PD and safety evaluation -Two regimens of ICP-022 (High dose QD and low dose BID) were designed for assessment of safety, as well as PK/PD profiles. The recommended dose of phase II clinical study will be determined according to the Part I results.

Part II: Dose expansion -Anti-tumor effects of ICP-022 in Chinese patients with R/R MCL will be evaluated in approximately 80 subjects. The recommended Phase 2 dose will be used in the Part II.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 75 years old
* Histologically confirmed mantle cell lymphoma (MCL), with either t(11;14) by cytogenetics and/or cyclin D1 overexpression by immunohistochemistry (IHC)
* Subjects with refractory or relapsed mantle cell lymphoma who has received at least 1 but no more than 4 prior therapies for MCL
* At least one measurable tumor of greater than 1.5 centimeter in long axis by contrast-enhanced CT/MRI
* ECOG performance status of 0-2
* Documented failure to achieve at least partial response (PR) or documented disease progression after response to, the most recent treatment regimen.
* Subjects who meet the following laboratory parameters:

  1. Absolute neutrophil count (ANC) ≥ 1.5×109/L Platelet count ≥ 75×109/L, independent of growth factor support within 7 days of the first dose with study drug, Hemoglobin ≥ 80 g/L; ANC ≥ 1.0×109/L, Platelet count ≥ 50×109/L if bone marrow involvement
  2. Total bilirubin ≤ 2× ULN; AST or ALT ≤ 2.5 ULN; Creatinine clearance ≥ 30ml/min; Amylase ≤ ULN and Lipase ≤ ULN
  3. International normalized ratio (INR) ≤ 1.5 ULN and activated partial thromboplastin time (APTT) ≤ 1.5 ULN
* Life expectancy ≥ 4 months
* Able to provide signed written informed consent

Exclusion Criteria:

* History of other active malignancies within 5 years of study entry, unless cured without evidence of relapse or metastasis
* Current or history of lymphoma involved central nervous system
* Prior corticosteroids (at dosages equivalent to prednisone > 20 mg/day) given with anti-neoplastic intent within 7 days, prior chemotherapy, targeted therapy, radiation therapy, or antibody based therapies or anti-cancer TCM within 4 weeks of the start of study drug.
* Non-hematological toxicity must recover to ≤ Grade 1 from prior anti-cancer therapy
* Current clinically significant cardiovascular disease including:

  * Any class 3 or 4 cardiac disease such as arrhythmia, congestive heart failure or myocardial infarction defined by the New York Heart Association Functional Classification, or left ventricular ejection fraction (LVEF) < 50%
  * Primary cardiomyopathy
  * Clinical significant QTc prolong history or QTc>470ms (female) QTc>450ms (male)
  * Uncontrolled hypertension
* Known active bleeding within 2 months of screening or currently taking anticoagulant/antiplatelet drugs
* Urine protein ≥ 2+ and quantitation ≥ 2g/24hours
* History of deep vein thrombosis or pulmonary embolism
* Disease significantly affecting gastrointestinal function such as dysphagia, chronic diarrhea, intestinal obstruction, or resection of the stomach
* Allogeneic stem cell transplant within 6 months prior to first dose of study drug or related active infection
* Major surgery within 6 weeks of screening, except for diagnostic test or vascular access setup
* Known active infection with HBV, HCV or HIV or any uncontrolled active systemic infection
* Any history of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonia, severe lung function impairment
* Prior exposure to a BTK inhibitor，BCR pathway ingibitor(such as PI3K, SYK) or BCL-2 kinase inhibitor
* Suitable and ready for allogeneic stem cell transplant
* Inability to comply with study procedures
* Drug abuser or alcoholics
* Lactating or pregnant women, or women who will not use contraception during the study and for 180 days after the last dose of study drug if sexually active and able to bear children
* Requires treatment with moderate or strong cytochrome P450 family 3, subfamily A (CYP3A) inhibitors or strong CYP3A inducers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-04-02 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | Up to 3 years
  The efficacy measured by overall response rate (ORR) in Part II according to the 2014 International Working Group NHL

SECONDARY OUTCOMES:
Occurrence of adverse events and serious adverse events according to NCI-CTCAE 4.03 grading criteria in Part I | Up to 3 years
  The safety of ICP-022 measured by the occurrence of adverse events and serious adverse events according to NCI-CTCAE 4.03 grading criteria in Part I
time to progression (TTP) | Up to 3 years
  The efficacy measured by time to progression (TTP) in Part II
progression free survival (PFS) | Up to 3 years
  The efficacy measured by progression free survival (PFS) in Part II
overall survival (OS) | Up to 3 years
  The efficacy measured by overall survival (OS) in Part II
Area under the concentration time curve up to the time "t" (AUC(0-t)) | up to 4 weeks
  Area under the concentration time curve up to the time "t" (AUC(0-t)) of ICP-022 will be measured and calculated with noncompartmental analysis using WinNonlin.
The percent of target occupancy | up to 4 weeks
  PBMC from individual subject before and after dosing will be collected and the target occupancy will be determined by ELISA. The percent of target occupancy will be compared descriptively.
Maximum plasma drug concentrations (Cmax) | up to 4 weeks
  Individual plasma concentrations of ICP-022 will be measured and Cmax will be calculated with noncompartmental analysis using WinNonlin.
Time of maximum plasma drug concentrations (Tmax) | up to 4 weeks
  Time of maximum plasma drug concentrations (Tmax) of ICP-022 will be recorded.
Apparent half-life for designated elimination phases (t½) | up to 4 weeks
  Apparent half-life for designated elimination phases (t½) of ICP-022 will be measured and calculated with noncompartmental analysis using WinNonlin.
Area under the concentration time curve up to the last data point above LOQ (AUC(last)) | up to 4 weeks
  Area under the concentration time curve up to the last data point above LOQ (AUC(last)) of ICP-022 will be measured and calculated with noncompartmental analysis using WinNonlin.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhu, PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (31):
- China (31):
  - Anhui Province Cancer Hospital, Hefei, Anhui
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Henan Tumor Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Tongji Hospital, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaojing
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - Qilu Hosptial of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Xin Hua Hospital Affiated to Shanghai Jiao Tong University School of Medicin, Shanghai, Shanghai Municipality
  - West China Hospital,Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhengjiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang

REFERENCES:
- [Derived] Deng LJ, Zhou KS, Liu LH, Zhang MZ, Li ZM, Ji CY, Xu W, Liu T, Xu B, Wang X, Gao SJ, Zhang HL, Hu Y, Li Y, Cheng Y, Yang HY, Cao JN, Zhu ZM, Hu JD, Zhang W, Jing HM, Ding KY, Zhang XY, Zhao RB, Zhang B, Tian YM, Song YP, Song YQ, Zhu J. Orelabrutinib for the treatment of relapsed or refractory MCL: a phase 1/2, open-label, multicenter, single-arm study. Blood Adv. 2023 Aug 22;7(16):4349-4357. doi: 10.1182/bloodadvances.2022009168. PMID 37078706